CLINICAL TRIAL: NCT06193369
Title: Digital Peer Navigation for Adolescents and Young Adults With Cancer: A Feasibility Study
Brief Title: Digital Peer Navigation for Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Young Adult Cancer Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-5552
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Breast Cancer; Testicular Cancer; Sarcoma
Keywords: Young Adults; Post-Treatment Cancer Survivorship; Digital Health; Patient Navigation; Peer Support; Patient Activation; Pilot RCT
MeSH Terms: conditions — Lymphoma; Breast Neoplasms; Testicular Neoplasms; Sarcoma; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention arm will the receive digital peer navigation intervention.
  Interventions: Behavioral: Digital Peer Navigation
- Waitlist Control (No Intervention): Participants assigned to the control arm will receive usual care. After completion of the study, they will have the option to receive the digital peer navigation intervention.

INTERVENTIONS:
Behavioral: Digital Peer Navigation — Participants in the intervention group will receive ongoing support from a trained peer navigator for 3 months after completing treatment for cancer. Participants will be matched through a digital app with a trained peer navigator who assesses needs and barriers to care, provides practical, informational, and emotional support, and empowers them to take a proactive role in their health. Patients will communicate with their peer navigator through digital direct messaging, videoconference or by telephone. Participants will also have access to a health resource library on the digital app that contains local and national resources about cancer.
  Arms: Intervention

SUMMARY:
Adolescents and young adults (AYA) diagnosed with cancer experience unique challenges after completing treatment and face distinct barriers to optimal care and support. These challenges include higher levels of symptom burden and treatment complications, interrupted education, careers and relationships, and financial hardship. AYA lack access to peers, relevant information and emotional support, and report gaps in care when dealing with these difficult challenges.

Digital peer navigation could help to address the needs of AYA and overcome barriers to care and support. The PI developed True North Peer Navigation (TrueNTH-PN), an evidence-based digital peer navigation program for men with prostate cancer and online peer navigator training course. The goal of this project is to adapt TrueNTH-PN for AYA and evaluate its feasibility to overcome barriers to care and support, and enhance patient activation among AYA during the challenging post-treatment phase.

In partnership with AYA cancer survivors, the Canadian Cancer Society, Young Adult Cancer Canada, a digital app design firm and technology provider, our cross-Canada team will: (1) Adapt and evaluate the usability of the TrueNTH-PN app for AYA; (2) Adapt and evaluate the effectiveness of the Peer Navigator Training Course for AYA; and (3) Determine the feasibility, acceptability and preliminary effectiveness of the new AYA-PN program among post-treatment AYA cancer survivors.

This project will produce an innovative solution to an important service gap in the lives of AYA with cancer. It has the potential to address the support needs of AYA, overcome barriers to care, and empower AYA to take proactive role in managing their health. In addition, it will give rise to AYA peer navigators with specialized skills, which could fill gaps in disrupted education and career paths, and help to attain future goals.

DETAILED DESCRIPTION:
Background: Adolescent and young adult (AYA) cancer survivors experience unique challenges and face distinct barriers to optimal post-treatment survivorship care and support which can impede their recovery. These include high levels of symptom burden and treatment-related complications, interrupted education, careers and relationships, and financial toxicity. AYA lack access to peers, relevant information and emotional support, and report gaps in care when dealing with these difficult challenges. Previous research has shown that patient navigation improves the timeliness of care and support, and reduces healthcare costs. Engaging trained volunteer cancer survivors as peer navigators minimizes resource requirements, is preferred by AYA over professional support, and benefits the navigator by improving their psychosocial health. The PI developed True North Peer Navigation (TrueNTH-PN), an evidence-based digital peer navigation program for men with prostate cancer and online competency-based peer navigator training course. Patients are matched through a digital app with a trained peer navigator who assesses needs and barriers to care, provides practical, informational, and emotional support, and empowers a proactive approach to health. TrueNTH-PN has been shown to be highly acceptable to prostate cancer patients and peer navigators, and associated with improvements in patient activation, social support and quality of life.

Aim: This study aims to adapt and evaluate a digital peer navigation program for AYA cancer survivors to overcome barriers to care and support, and enhance patient activation during the post-treatment survivorship phase.

Specific Objectives: This 3-phase project will: (1) Adapt and evaluate the usability of the TrueNTH-PN app for AYA; (2) Adapt and evaluate the effectiveness of TrueNTH-PN peer navigator training course for AYA; and (3) Determine the feasibility, acceptability and preliminary effectiveness of the new AYA peer navigation program (AYA-PN).

Methods: We will adopt an iKT approach with patients, Canadian Cancer Society and Young Adult Cancer Canada as partners, along with a digital app design firm and technology provider. For objective 1, informed by Barrera and Castro's cultural adaptation framework and user-centred design, we will engage AYA in a critical assessment of the existing TrueNTH-PN app to identify areas in need of adaptation for AYA, co-design content and processes adaptations, and conduct user-testing. For objective 2, we will tailor and validate the relevance of the course content for AYA; recruit, screen and train 20 AYA cancer survivors to be peer navigators; and informed by the Kirkpatrick training program framework, evaluate the training course using pre-post questionnaires to assess knowledge and self-efficacy for navigator competencies. For objective 3, we will conduct a pilot RCT of the new AYA-PN program compared to wait list control with an embedded process evaluation to determine: 1) feasibility; 2) acceptability; and 3) preliminary effectiveness on patent activation, supportive care needs, quality of life, anxiety/depression, social support and post-traumatic growth. One hundred thirty eight AYA (n=69 per arm) will be recruited after completing treatment. Outcomes will be assessed at baseline (T0) and 3-months (T1). In addition, we will evaluate patient-navigator interactions, app usage, and cost-effectiveness, and conduct semi-structured interviews with patients and navigators informed by the Consolidated Framework for Implementation Research to capture experiences, explore mechanisms of action and identify implementation barriers and facilitators.

Significance: This study will produce an innovative solution to an important service gap in the lives of AYA with cancer. It is highly aligned with the CCS priority in AYA survivorship care, the Pan-Canadian Cancer Survivorship Research Agenda, and the SPOR mandate to make research more responsive to the needs of Canadians.

ELIGIBILITY:
Inclusion criteria:

1. Are 18-40 years old;
2. Were diagnosed with breast or testicular cancer, lymphoma or sarcoma between the ages of 15-39 years old;
3. Have completed therapy within the last 12 months;
4. Are comfortable using the internet;
5. Have an active email address OR are willing to create one;
6. Able to read and speak English.

Exclusion criteria:

1. Have metastatic disease or are receiving palliative end-of-life care;
2. Are not willing to be randomized.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient activation | 0, 3 months
  The primary outcome will be change in Patient Activation from baseline to 3 months. Patient Activation will be measured using the Patient Activation Measure (PAM). Higher scores represent a better outcome.

SECONDARY OUTCOMES:
Health utility | 0, 3 months
  Health utility will be measured with the EQ-5D.
Supportive care needs | 0, 3 months
  Supportive care needs will be measured with the Supportive Care Needs Survey (SCNS-SF34).
Anxiety | 0, 3 months
  Anxiety will be measured with the Generalized Anxiety Disorder scale (GAD-7).
Depression | 0, 3 months
  Depression will be measured with the Patient Health Questionnaire (PHQ-9).
Social support | 0, 3 months
  Social support will be measured with the ENRICHD Social Support Instrument (ESSI).

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Bender, PhD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No